CLINICAL TRIAL: NCT06479538
Title: Comparative Effects of Post Isometric Relaxation and Post Facilitation Stretching on Pain, Rom and Functional Disability Among Young Fast Bowlers With Quadratus Lumborum Tightness
Brief Title: Effects of Post Isometric Relaxation and Post Facilitation Stretching on Young Fast Bowlers
Acronym: (PIR)(PFS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0489 AMAMA
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
Keywords: Back pain; muscle energy technique; Quadratus lumborum; visual analogue pain scale; disability
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 17 participants will be in experimental group A giving them Post isometric relaxation of Quadratus lumborum for four weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Post isometric relaxation
- Group B (Experimental): 17 participants will be in experimental group B giving them Post facilitation stretching of Quadratus lumborum for four weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Post facilitation stretching

INTERVENTIONS:
Other: Post isometric relaxation — 17 participants will be in experimental group A giving them Post isometric relaxation of Quadratus lumborum for four weeks, measuring all values before giving them protocol and after protocol.
  Arms: Group A
Other: Post facilitation stretching — 17 participants will be in experimental group A giving them Post facilitation stretching of Quadratus lumborum for four weeks, measuring all values before giving them protocol and after protocol.
  Arms: Group B

SUMMARY:
The quadratus lumborum muscle exhibited the highest degree of asymmetry in fast bowlers with low back pain, the identification and correction of this asymmetry is always of interest. Fast bowlers in cricket are more likely to experience non-contact LBP if they use improper technique, prepare less physically, ball too hard, or take on an excessive workload. The quadratus lumborum muscle exhibited the highest degree of asymmetry in fast bowlers with low back pain due to extreme side flexion at non-dominant side and hence results in QL tightness at that side.

The study design will be a Randomized Controlled Trial. This study will be conducted in Pakistan Sports Board (PSB) Lahore. The study will be completed within the time duration of eight to ten months after the approval of the synopsis. The sample size will be 34 subjects. Non-probability convenient sampling technique will be used to recruit the individuals for the study. Then randomization will be done by lottery method to divide the individuals into 2 treatment groups. The experimental group A will be given Post isometric relaxation for 20 minutes for 4 weeks (four times per week) on the other hand experimental group B will receive Post facilitation stretching and after that measure their pre-post values on SPSS. Pain will be measured with VAS, range of motion with inclinometer and functional disability with athlete's disability index questionnaire. In this study, it will be aimed to examine the comparative effects of both techniques that affect pain, range of motion and functional disability with quadratus lumborum tightness in young fast bowlers.

DETAILED DESCRIPTION:
The main objective of this study is to apply post isometric relaxation and post facilitation stretching techniques and to compare the results to identify their influence on pain, range of motion and functional disability on quadratus lumborum tightness in young fast bowlers.

ELIGIBILITY:
Inclusion Criteria:

* Age15-19years
* both male and female fast bowlers
* passive pelvic transverse gliding test for Quadratus lumborum tightness +ve
* Low back pain > 6 weeks
* Training sessions of at least 3 days/week

Exclusion Criteria:

1. Congenital causes (Spina bifida, Scoliosis, Spondylosis, Spondylolisthesis)
2. Traumatic cause

   * Prolapsed intervertebral disc
   * fracture of vertebral column
3. Inflammatory cause

   * Ankylosing spondylosis
   * Pott's spine
4. Neoplastic cause

   * Benign
   * Malignant
5. Radiculopathy
6. Any spinal surgery
7. Gynecological cause

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Participants are asked to rate their low back pain from 0 to 10. It is a psychometric response scale that is used in Questionnaires. It is used to measure the perceived Pain intensity. The numbers are given from a range of 0-10 classifying as mild, moderate and severe pain. (21)
Inclinometer | 4 weeks
  Range of motion of trunk lateral flexion is measured by inclinometer. An instrument used to measure an object's angles of elevation/depression and slope/tilt with regard to gravity is called an inclinometer, also known as a clinometer. The resultant measurement is expressed as a percentage with respect to a level zero plane or as an angular measurement (degrees, minutes, seconds, etc.) (22)
Athletes Disability Index Questionnaire | 4 weeks
  The ADI is a self-administered questionnaire designed to evaluate athletes' disabilities related to low back pain. In addition to limitations in activities of daily life, the ADI also covers functional disabilities in sports and exercise. The 12 questions in the ADI cover a variety of topics, including the degree of pain, stretching, strengthening, and weight training exercises, technical skills specific to a sport, rotational back movements and direction changes, fear of pain or (re)injury, sitting, walking, recreational activities, sexual activity, sleep, and self-care (23)

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punajb, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jairakdee Y, Chansirinukor W, Sitti T. Effect of releasing quadratus lumborum muscle on hip and knee muscle length in asymptomatic individuals. J Bodyw Mov Ther. 2021 Apr;26:542-547. doi: 10.1016/j.jbmt.2020.11.008. Epub 2020 Nov 7. PMID 33992295
- [Background] Ranson C, Burnett A, O'Sullivan P, Batt M, Kerslake R. The lumbar paraspinal muscle morphometry of fast bowlers in cricket. Clin J Sport Med. 2008 Jan;18(1):31-7. doi: 10.1097/JSM.0b013e3181618aa2. PMID 18185036
- [Background] Hides J, Stanton W, Freke M, Wilson S, McMahon S, Richardson C. MRI study of the size, symmetry and function of the trunk muscles among elite cricketers with and without low back pain. Br J Sports Med. 2008 Oct;42(10):809-13. doi: 10.1136/bjsm.2007.044024. Epub 2007 Dec 7. PMID 18065440
- [Background] Senington B, Lee RY, Williams JM. Biomechanical risk factors of lower back pain in cricket fast bowlers using inertial measurement units: a prospective and retrospective investigation. BMJ Open Sport Exerc Med. 2020 Aug 13;6(1):e000818. doi: 10.1136/bmjsem-2020-000818. eCollection 2020. PMID 32843992
- [Background] Kountouris A, Portus M, Cook J. Cricket fast bowlers without low back pain have larger quadratus lumborum asymmetry than injured bowlers. Clin J Sport Med. 2013 Jul;23(4):300-4. doi: 10.1097/JSM.0b013e318280ac88. PMID 23377354
- [Background] Forrest MRL, Hebert JJ, Scott BR, Dempsey AR. Exercise-based injury prevention for community-level adolescent cricket pace bowlers: A cluster-randomised controlled trial. J Sci Med Sport. 2020 May;23(5):475-480. doi: 10.1016/j.jsams.2019.12.009. Epub 2019 Dec 17. PMID 31874733
- [Background] Eftekharsadat B, Fasaie N, Golalizadeh D, Babaei-Ghazani A, Jahanjou F, Eslampoor Y, Dolatkhah N. Comparison of efficacy of corticosteroid injection versus extracorporeal shock wave therapy on inferior trigger points in the quadratus lumborum muscle: a randomized clinical trial. BMC Musculoskelet Disord. 2020 Oct 19;21(1):695. doi: 10.1186/s12891-020-03714-3. PMID 33076888
- [Background] Fraeulin L, Holzgreve F, Brinkbaumer M, Dziuba A, Friebe D, Klemz S, Schmitt M, Theis A AL, Tenberg S, van Mark A, Maurer-Grubinger C, Ohlendorf D. Intra- and inter-rater reliability of joint range of motion tests using tape measure, digital inclinometer and inertial motion capturing. PLoS One. 2020 Dec 10;15(12):e0243646. doi: 10.1371/journal.pone.0243646. eCollection 2020. PMID 33301541
- [Background] Noormohammadpour P, Hosseini Khezri A, Farahbakhsh F, Mansournia MA, Smuck M, Kordi R. Reliability and Validity of Athletes Disability Index Questionnaire. Clin J Sport Med. 2018 Mar;28(2):159-167. doi: 10.1097/JSM.0000000000000414. PMID 28107217